CLINICAL TRIAL: NCT04996810
Title: A Randomized, Double-blinded, Active Comparator, Single-dose, Phase I/II Trial to Evaluate the Safety and Efficacy of Treatment With PROTOXIN as Compared to BOTOX® in Adult Subjects Who Need Improvement of Moderate or Severe Glabellar Lines
Brief Title: The Safety and Efficacy Study of PROTOXIN in Subjects With Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Protox Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PT_BTA_P1_20
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Glabellar Frown Lines
Keywords: Glabellar Lines; Botulinum toxin; Botulinum toxin type A
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROTOXIN (Phase I/II) (Experimental): PROTOXIN will be injected to 5 glabellar lines (Each 4U/0.1mL, Total 20U/0.5mL).
  Interventions: Biological: PROTOXIN
- Botox® (Phase II) (Active Comparator): Botox® will be injected to 5 glabellar lines (Each 4U/0.1mL, Total 20U/0.5mL).
  Interventions: Biological: Botox®

INTERVENTIONS:
Biological: PROTOXIN — Botulinum toxin Type A
  Arms: PROTOXIN (Phase I/II)
Biological: Botox® — Botulinum toxin Type A
  Arms: Botox® (Phase II)

SUMMARY:
This study will be conducted in Phase I/II clinical trials. In Phase I, subjects with moderate to severe glabellar lines are enrolled and those who are judged to be eligible for this study will be injected with the "PROTOXIN" at a total of 20U(4U/0.1mL each) in five sites of the glabellar lines. Safety is assessed after 12 weeks. In Phase II, subjects with moderate to severe glabellar lines are enrolled and will be injected the "PROTOXIN" or the "BOTOX®" at a total of 20U(4U/0.1mL each)in five sites of the glabellar lines. Thereafter, efficacy and safety are assessed by comparing with BOTOX®.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 19 to 65 years old
* Subjects attaining ≥grade 2 (moderate) in the investigator's rating of the severity of glabellar lines at maximum frown
* Fertile women who have properly agreed to contraception during the clinical trial period
* Subjects who voluntarily sign the informed consent

Exclusion Criteria:

* Subjects who answered 'Yes' any of the C-SSRS questions (only Phase I)
* Subjects with the general neuromuscular synaptic disorder(e.g. Myasthenia gravis, Lambert-Eaton syndrome)
* Subjects who suffer from muscle weakness or paralysis in the forehead area
* Subjects with infection, skin disorders, or scars at the glabellar region.
* Subjects with noticeable facial asymmetry
* Subjects with allergy or hypersensitivity to the botulinum toxin or their components
* Subjects who have taken Anti-Coagulant, Anti-Platelet agent, Aspirin and NSAIDs within 7 days prior to administration of the investigational drug
* Subjects who were injected facial with botulinum toxin within the past 6 months or whose dose exceeds 200 U for the whole body
* Subjects with previous treatment of Face Lifting, Permanent Implant, and/or Filler in the glabellar region
* Subjects who are participating in other clinical trials or have participated in other clinical trials within 4 weeks of the screening date.
* A history of drug or alcohol abuse
* Fertile women and men who have plans to conceive during pregnancy, breastfeeding and clinical trials or who do not agree to appropriate contraception
* Subjects who are not eligible for this study based on the judgment of an investigator

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Evaluate the Number of subjects with treatment-related adverse events as assessed by CTCAE Version 5.0 (Phase I) | 12 weeks after the injection
Glabellar line improvement rate confirmed with investigator's assessment (Phase II) | 4 weeks after the injection

SECONDARY OUTCOMES:
Glabellar line improvement rate confirmed with investigator's assessment (Phase II) | 4, 8, 12 weeks after the injection
Glabellar line improvement rate confirmed by subject' satisfaction assessment (Phase II) | 4, 8, 12 weeks after the injection
Evaluate the Number of subjects with treatment-related adverse events as assessed by CTCAE Version 5.0 (Phase II) | 12 weeks after the injection

CONTACTS AND LOCATIONS:
Overall Officials: Beomjoon Kim, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (2):
- South Korea (2):
  - Chung-Ang University Hospital, Seoul
  - Nowon Eulji Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No